CLINICAL TRIAL: NCT06397898
Title: NOVasure Endometrial Ablation Pre-, Peri- and Postprocedural Patient's EXperiences and Satisfaction for Women With Heavy Menstrual Bleeding (the NOVEX Trial): A Qualitative Questionnaire Pilot-study
Brief Title: NOVasure EXpierences (NOVEX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Nadia Dkhissi, N.Dkhissi, BA in Medicine, Principal Investigator, Maxima Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N21.091
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Abnormal Uterine Bleeding
Keywords: endometrial ablation
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Intervention Model Description: Randomized-controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (video) (Experimental): group that viewed an educational video before Novasure treatment
  Interventions: Other: Educational video
- Control group (no video) (No Intervention): group that did not view an educational video before Novasure treatment

INTERVENTIONS:
Other: Educational video — Viewing an educational video before Novasure treatment
  Arms: Intervention group (video)

SUMMARY:
Heavy menstrual bleeding (HMB) affects approximately one in four women and imposes considerable social, emotional, physical and economic burdens. Despite various treatment options available, endometrial ablation (Novasure) has emerged as a promising solution, with documented efficacy and high patient satisfaction rates. In the context of peri- and postoperative pain, research has reported that patients experienced less pain during the Novasure endometrial ablation procedure in comparison with two other systems. Moreover, postoperative pain rates were lower in patients treated with Novasure compared to another endometrial ablation device (ThermaChoice system).

Nonetheless, it remains unclear how patients in detail experience the Novasure treatment. It is not clear which factors contribute to either a positive or a negative experience. Moreover, it is unknown if women wish more education before the procedure in order to feel well prepared for the procedure and possible post-procedural symptoms. Therefore, we want to investigate how women with heavy menstrual bleeding experience education about endometrial ablation (Novasure) treatment, the procedure itself and short-term care after treatment.

In this randomized-controlled pilot study, the aim is :

1. To determine if educational videos that show experiences from women with HMB that were treated with Novasure endometrial ablation affect preoperative anxiety.
2. To assess if educational videos have an effect on preoperative need for information
3. To explore Novasure pre-, peri- and postoperative patient experiences
4. To define positive and negative factors related to Novasure endometrial ablation
5. To gain insight in factors that could improve patient satisfaction before, during and after Novasure endometrial ablation and to evaluate the educational videos.

DETAILED DESCRIPTION:
Procedure:

Subjects will be recruited from the outpatient clinic from Máxima Medical Center Eindhoven and Veldhoven. Patients presenting with heavy menstrual bleeding and scheduled for endometrial ablation (Novasure) between March 2022 and April 2024 were approached for study participation either by email, phone call, or in-person during their clinic visit. Upon expressing interest, patients will be provided with detailed information about the study and asked to sign an informed consent form. Patients were randomized in an alternating order and 1:1 ratio.

Subsequently, after randomization, the participants will be sent a secure email containing the link to the educational videos. Patients will watch the educational videos 1-7 days before their Novasure treatment.On the day of treatment, before undergoing the Novasure procedure, patients will complete the Visual Analogue Scale for Anxiety (VAS-A) and Amsterdam Preoperative Anxiety and Information Scale (APAIS).

Two days post-treatment, the participants will receive a questionnaire via email through Research Manager. This questionnaire will encompass inquiries regarding demographics, patient characteristics, treatment-related positive and negative factors, improvement of care, and patient satisfaction.

Two groups will complete the questionnaires: one group that viewed an educational video before Novasure treatment and a control group that did not view the video. Both groups receive the same treatment (Novasure), with the only difference being the addition of the educational video as part of pre-procedural preparation, as both groups receive information from the gynecologist about the procedure. Additionally, patients have access to further information online or in brochures. Therefore, conducting this study raises no ethical concerns.

The researchers conducted a power calculation using G*Power 3 to determine the sample size for the questionnaire research. Based on this calculation, considering a pilot study and prior research suggesting a minimum of 12 patients per group, the aim was to include 16 patients per group (total 32 patients).

Data will be analyzed by an intention-to-treat analysis. Frequencies and percentages for general characteristics will be determined. The mean plus standard deviation of VAS-A, APAIS anxiety and need to obtain information scores, and other scale variables will be calculated. Mann-Whitney U tests will be used to assess group differences for VAS-A, APAIS, and scale variables. A p<0.05 will be considered statistically significant. Descriptive statistics will be used to compute frequencies and corresponding percentages for nominal and ordinal variables.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for heavy menstrual bleeding with endometrial ablation (Novasure) between the period of March 2022 and May 2024
* Age 18-60 years
* No wish to conceive a pregnancy in the future

Exclusion Criteria:

* No written informed consent for the interview and distribution of the final educational video which includes relevant pieces from the interview
* Patients that do not speak, read and/or write in Dutch
* Pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | Patients fill out the VAS-A form in the hospital shortly before the procedure.
  Preoperative anxiety, measured by the Visual Analogue Scale for Anxiety (VAS-A), is the primary outcome. The VAS is a 100 mm line, and patients are asked to mark their anxiety level on this line. The left end of the line represents "no anxiety," and the right end represents "worst imaginable anxiety." VAS-A is noted in millimeters. Patients fill out the VAS-A form in the hospital shortly before the procedure.

SECONDARY OUTCOMES:
Preoperative anxiety and the need to obtain information about the procedure and anesthesia. | Together with the VAS-A, the APAIS is filled out by patients shortly before the procedure.
  Measured by the Amsterdam Preoperative Anxiety and Information Scale (APAIS) . Anxiety scores are calculated by adding up the scores of questions 1, 2, 4, and 5. Patients with an anxiety score of ≥11 are considered anxious. Information need scores are calculated by adding up the scores of question 3 and 6. A score between 2-4 represents no to little need to obtain information, a score between 5-7 represents an average need to obtain information, and a score between 8-10 represents a high need to obtain information about the procedure and anesthesia.
To asses patient experiences and satisfaction, related to endometrial ablation. | two days after post-treatment
  Patients will fill in an online questionnaire, including questions about demographics, patient characteristics, treatment-related positive and negative factors, improvement of care, and patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Máxima Medical Center, Veldhoven, North Brabant, Netherlands